CLINICAL TRIAL: NCT04316364
Title: A Randomized, Double-Blind, Multicenter, Phase Ib/III Clinical Study on PD-L1 Monoclonal Antibody SHR-1316 or Placebo in Combination With Chemotherapy as Perioperative Treatment of Resectable Stage II or III Non-Small Cell Lung Cancer
Brief Title: A Trial of SHR-1316/Placebo in Combination With Chemotherapy in Patients With Resectable NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1316-III-303
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): Neoadjuvant setting: Drug: SHR-1316 and carboplatin and Paclitaxel (Albumin Bound) 3 cycles; Adjuvant setting: Drug: SHR-1316 up to 16 cycles
  Interventions: Drug: SHR-1316、Paclitaxel (Albumin Bound)、Carboplatin
- Treatment group B (Experimental): Neoadjuvant setting: Drug: SHR-1316 and platinum-based dual chemotherapy 3 cycles; Adjuvant setting: Drug: SHR-1316 up to 16 cycles
  Interventions: Drug: SHR-1316、Chemotherapeutic
- Treatment group C (Placebo Comparator): Neoadjuvant setting: Drug: Placebo and platinum-based dual chemotherapy 3 cycles; Adjuvant setting: Drug: Placebo up to 16 cycles
  Interventions: Drug: Placebo、Chemotherapeutic

INTERVENTIONS:
Drug: SHR-1316、Paclitaxel (Albumin Bound)、Carboplatin — Drug: SHR-1316, an engineered anti-PD-L1 antibody will be administered as intravenous (IV) infusion on Day 1 of each 21-day cycle Drug: Paclitaxel (Albumin Bound) will be administered intravenously on Day 1,8,15 of each 21-day cycle Drug: Carboplatin will be administered intravenously on Day 1 of each 21-day cycle
  Arms: Treatment group A
Drug: SHR-1316、Chemotherapeutic — Drug: SHR-1316, an engineered anti-PD-L1 antibody will be administered as intravenous (IV) infusion on Day 1 of each 21-day cycle Drug: Chemotherapeutic drugs will be administered on Day 1 of each 21day cycle, if applicable, they will also be administered on Day 8 and/or Day 15 according to the drug package insert
  Arms: Treatment group B
Drug: Placebo、Chemotherapeutic — Drug: Placebo, will be administered as intravenous (IV) infusion on Day 1 of each 21-day cycle Drug: Chemotherapeutic drugs will be administered on Day 1 of each 21day cycle, if applicable, they will also be administered on Day 8 and/or Day 15 according to the drug package insert
  Arms: Treatment group C

SUMMARY:
This trial is designed to evaluate the efficacy, safety and immunogenicity of neoadjuvant treatment with monoclonal antibody SHR-1316 or placebo in combination with platinum doublet chemotherapy in participants with resectable Stage II, IIIA, or selected IIIB non-small cell lung cancer (NSCLC) followed by adjuvant SHR-1316 or placebo and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Have previously untreated, pathologically confirmed resectable Stage II, IIIA, or Selected IIIB NSCLC. Staging should be based on the 8th edition of the AJCC/UICC staging system
* Evaluation by an attending thoracic surgeon to confirm eligibility for an R0 resection with curative intent
* Adequate tumor tissue sample blocks for central programmed death-ligand 1 (PD-L1) testing
* Measurable disease as defined by RECIST v1.1
* Adequate organ function
* Women of childbearing age without sterilizing or male, must agree to use contraception or practice abstinence at least 180 days after the last dose of study treatment

Exclusion Criteria:

* Any previous systematic anti-cancer therapy for lung cancer
* With active, known or suspected autoimmune disease of autoimmune disease
* Malignancies other than NSCLC within 5 years prior to randomization
* Has or suspected has a history of pneumonitis /interstitial lung disease or any serve lung diseases which will influence the examination of lung function
* Significant history of cardiovascular and cerebrovascular disease
* Significant haemorrhagic disease
* Has an arteriovenous thrombotic events
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known active Hepatitis B or Hepatitis C
* Allergic to monoclonal antibodies or other protein drugs
* Allergic to the intervention regimens
* Pregnant or lactating women
* Has known psychiatric or substance abuse disorders
* Confirmed COVID-19 infection or suspected COVID-19 infection or close contact with a person with known or suspected COVID-19 infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | At time of surgery
Event free survival (EFS) | Approximately 66 months

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 96 months
Pathology complete response (pCR) | At time of surgery
Objective response rate (ORR) | prior to surgery
Disease-Free Survival (DFS) | Approximately 66 months

CONTACTS AND LOCATIONS:
Overall Officials: YILONG WU, M.D, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - JiangSu Cancer Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang